CLINICAL TRIAL: NCT03194243
Title: Pathway and Urgent caRe of Dyspneic Patient at the Emergency Department in LorrainE District
Brief Title: Pathway and Urgent caRe of Dyspneic Patient at the Emergency Department in LorrainE District (PURPLE)
Acronym: PURPLE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-A01877-44
Record Dates: First submitted 2017-05-29; First posted 2017-06-21 (Actual); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Acute Dyspnea
Keywords: acute dyspnea; acute heart failure; emergency
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients admitted for acute dyspnea: Patients admitted for acute dyspnea in the emergency department

SUMMARY:
This is an observational prospective multicenter study of patients admitted for acute dyspnea in an emergency department of the participating centers in the Lorraine district.

The primary objective is to assess the outcome of this population according to the cause of acute dyspnea as well as identify the predictors of this outcome, both overall and according to each acute dyspnea cause.

DETAILED DESCRIPTION:
This observational prospective multicenter study will be conducted using data from electronic medical records, acquired as part of usual care, in patients admitted for acute dyspnea in the emergency department. Clinical, treatment, laboratory and imaging data acquired during the hospitalization (in the emergency department and in the department that admitted the patients following the emergency department stay) will be collected.

Vital status will be recorded at 30 days and 1 year post-admission.

ELIGIBILITY:
Inclusion Criteria:

* Men or women > or = 18 years.
* Patients with acute dyspnea admitted for acute dyspnea in the emergency department.
* Patient informed.

Exclusion Criteria:

* Cardiorespiratory arrest.
* Patient having expressed his or her opposition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute dyspnea and treated in an emergency department of the participating centers in the Lorraine district.
Sampling Method: Non-Probability Sample
Enrollment: 75000 (Estimated)
Dates: Start 2017-10-05 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | From emergency admission for acute dyspnea up until 1 year

SECONDARY OUTCOMES:
Demographic data | through hospital stay, an average of 10 days
Clinical data | through hospital stay, an average of 10 days
Treatment data | through hospital stay, an average of 10 days
Laboratory data | through hospital stay, an average of 10 days
Imaging data | through hospital stay, an average of 10 days
Duration of hospitalization | At final discharge, an average of 10 days after admission
  including emergency stay and conventional hospitalization
Initial diagnosis in the emergency department | At admission
Final diagnosis of the initial hospitalization stay | At final discharge, an average of 10 days after admission
Brain Natriuretic Peptide | Through hospital stay, an average of 10 days
Estimated glomerular function rate | Through hospital stay, an average of 10 days
Estimated plasma volume | Through hospital stay, an average of 10 days
Liver biological biomarkers | Through hospital stay, an average of 10 days
Urea | Through hospital stay, an average of 10 days
Use of non-invasive ventilation | Through hospital stay, an average of 10 days
Time of use of non-invasive ventilation | Through hospital stay, an average of 10 days
Use of diuretics | Through hospital stay, an average of 10 days
Time of use of diuretics | Through hospital stay, an average of 10 days
Use of nitrates | Through hospital stay, an average of 10 days
Time of use of nitrates | Through hospital stay, an average of 10 days
Department type admitting the patient following emergency management | Through hospital stay, an average of 10 days
  intensive care unit, cardiology, cardiac intensive care unit, other ...
All cause in-hospital mortality | At final discharge, an average of 10 days after admission

CONTACTS AND LOCATIONS:
Overall Officials: Tahar CHOUIHED, MD, Principal Investigator — Central Hospital, Nancy, France; Nicolas GIRERD, MD,PhD, Principal Investigator — Central Hospital, Nancy, France
Locations (9):
- France (9):
  - CH EPINAL - Service des Urgences, Épinal, Lorraine
  - CH Marie-Madeleine FORBACH - Service des Urgences, Forbach, Lorraine
  - CH LUNEVILLE - Service des Urgences, Lunéville, Lorraine
  - CHR METZ-THIONVILLE- Hôpital de Mercy- Service des Urgences, Metz, Lorraine
  - CHRU Nancy - Service des Urgences, Nancy, Lorraine
  - CH PONT A MOUSSON- Service des Urgences, Pont-à-Mousson, Lorraine
  - CH REMIREMONT - Service des Urgences, Remiremont, Lorraine
  - CH SAINT-DIE-DES-VOSGES - Service des Urgences, Saint-Dié, Lorraine
  - CHR METZ-THIONVILLE- Hôpital Bel-Air- Service des Urgences, Thionville, Lorraine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buessler A, Chouihed T, Duarte K, Bassand A, Huot-Marchand M, Gottwalles Y, Penine A, Andre E, Nace L, Jaeger D, Kobayashi M, Coiro S, Rossignol P, Girerd N. Accuracy of Several Lung Ultrasound Methods for the Diagnosis of Acute Heart Failure in the ED: A Multicenter Prospective Study. Chest. 2020 Jan;157(1):99-110. doi: 10.1016/j.chest.2019.07.017. Epub 2019 Aug 2. PMID 31381880